CLINICAL TRIAL: NCT00548691
Title: A Multi-center, Randomized Controlled Study to Investigate the Safety and Tolerability of IV Ferric Carboxymaltose (FCM) vs Standard Medical Care in Treating Iron Deficiency Anemia in Chronic Kidney Disease Patients
Brief Title: Safety and Tolerability of FCM vs Standard of Care in Treating Iron Deficiency Anemia in Chronic Kidney Disease Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: American Regent, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1VIT07018
Record Dates: First submitted 2007-10-22; First posted 2007-10-24 (Estimated); Results first posted 2015-05-13 (Estimated); Last update posted 2018-02-20 (Actual); Status verified 2018-01

CONDITIONS: Anemia
MeSH Terms: conditions — Anemia | interventions — ferric carboxymaltose

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ferric Carboxymaltose (FCM) (Experimental): Subjects received an undiluted dose of iron as FCM IV (15 mg/kg up to a maximum of 1000 mg) or subjects received 200 mg of FCM IV push undiluted directly into the venous line of the dialyzer.
  Interventions: Drug: Ferric Carboxymaltose
- Standard Medical Care (SMC) (Active Comparator): SMC for IDA (as determined by the Investigator) for treating CKD related anemia.
  Interventions: Drug: Standard Medical Care (SMC)

INTERVENTIONS:
Drug: Ferric Carboxymaltose
  Arms: Ferric Carboxymaltose (FCM)
Drug: Standard Medical Care (SMC)
  Arms: Standard Medical Care (SMC)

SUMMARY:
The Objective of this study is to study the safety of FCM in patients with anemia caused by chronic kidney failure

ELIGIBILITY:
Inclusion Criteria:

* Male or Female 18 to 85 years of age
* NDD-CKD Patients
* TSAT </= 25%
* Hgb </= 11.5
* Ferritin </= 300
* HD-CKD Patients
* TSAT </= 30%
* Hgb </= 12
* Ferritin </= 500

Exclusion Criteria:

* Previous participation in a FCM trial
* Known Hypersensitivity to FCM
* History of anemia other that anemia due to chronic renal failure
* Current history of GI bleeding
* Received IV Iron within the last 30 Days
* Anticipated need for surgery
* Malignancy history
* AST or ALT greater than normal
* Received an investigational drug within 30 days of screening
* Pregnant or sexually active females who are not willing to use an effective form of birth control

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 513 (Actual)
Dates: Start 2007-10; Primary Completion 2009-01 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Luitpold Pharmaceuticals, Norristown, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Hospitals and medical clinics
Period: Overall Study
Arm/Group | Ferric Carboxymaltose (FCM) | Standard Medical Care (SMC)
Started | 258 | 259
Completed | 251 | 250
Not Completed | 7 | 9

BASELINE CHARACTERISTICS:
Population: Safety population - of the 517 total subjects randomized, 4 subjects randomized to FCM were discontinued from the study prior to dosing due to selection critirea/study compliance (3 subjects) and subject request (1 subject)
Groups:
- Total: Total of all reporting groups
Arm/Group | Ferric Carboxymaltose (FCM) | Standard Medical Care (SMC) | Total
Number analyzed (Participants) | 254 | 259 | 513
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 127 | 126 | 253
  >=65 years | 127 | 133 | 260
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.5 (12.81) | 63.1 (12.11) | 62.8 (12.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 159 | 153 | 312
  Male | 95 | 106 | 201
Region of Enrollment [Number; unit: participants]
  United States | 254 | 259 | 513

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Treatment-emergent Serious Adverse Events (SAE's)
Time Frame: from Day 0 through 30 days after the last dose of study drug
Measure: Number; unit: participants
Arm/Group | Ferric Carboxymaltose (FCM) | Standard Medical Care (SMC)
Number analyzed (Participants) | 254 | 259
participants | 11 | 36

ADVERSE EVENTS:
Time Frame: 1 year and 2 months
Arm/Group | Ferric Carboxymaltose (FCM) | Standard Medical Care (SMC)
Serious Adverse Events (participants affected / at risk) | 11/254 | 36/259
Other Adverse Events (participants affected / at risk) | 0/254 | 0/259
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ferric Carboxymaltose (FCM) (N=254) | Standard Medical Care (SMC) (N=259)
Atrial flutter (Cardiac disorders) | 1 | 1
Hypovolemia (Metabolism and nutrition disorders) | 0 | 3
Osteomyelitis (Infections and infestations) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 3
Sepsis (Infections and infestations) | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 1
Ascities (Gastrointestinal disorders) | 0 | 1
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 2
Localized infection (Infections and infestations) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Catheter related complication (General disorders) | 0 | 1
Ventricular fibrillation (Cardiac disorders) | 0 | 1
Vitreous hemorrhage (Eye disorders) | 1 | 0
Thromboembolic stroke (Nervous system disorders) | 0 | 1
Clostridial infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1
Azotemia (Renal and urinary disorders) | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 1
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 0
Anemia (Blood and lymphatic system disorders) | 0 | 2
Constipation (Gastrointestinal disorders) | 0 | 1
Renal failure acute (Renal and urinary disorders) | 0 | 1
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Angina pectoris (Cardiac disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1
Urosepsis (Infections and infestations) | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0
Catheter sepsis (Infections and infestations) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less